CLINICAL TRIAL: NCT06896318
Title: Virtual Reality-Supported Cardiac Rehabilitation: Psychological, Functional, and Physiological Perspectives
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Jan Dlugosz University in Czestochowa (Other); Provincial Specialist Hospital of the Blessed Virgin Mary in Częstochowa (Unknown)
Responsible Party: Principal Investigator, Błażej Cieślik, Principal Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54/2024
Record Dates: First submitted 2025-02-07; First posted 2025-03-26 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Coronary Arterial Disease (CAD); Myocardial Disease; Heart Disease
Keywords: virtual reality; relaxation; cardiac rehabilitation; kinesiophobia; stress; depression; new technologies; heart disease
MeSH Terms: conditions — Cardiovascular Diseases; Cardiomyopathies; Heart Diseases; Kinesiophobia; Depression | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Group (Experimental): Cardiac rehabilitation supplemented by VR therapy
  Interventions: Device: Virtual Reality Therapy; Behavioral: Cardiac rehabilitation
- Control Group (Active Comparator): Conventional cardiac rehabilitation
  Interventions: Behavioral: Cardiac rehabilitation

INTERVENTIONS:
Device: Virtual Reality Therapy — 8 sessions of VR therapy (each of them 20 minutes long). As a virtual reality source, VR TierOne device (Stolgraf®) were used. Thanks to using head mounted display and the phenomenon of total immersion VR therapy provides an intense visual, auditory and kinesthetic stimulation. It can have a calming and mood-improving effect or help the patients recognize their psychological resources and motivate to the rehabilitation process. In the virtual therapeutic garden there are a rich set of symbols and metaphors based on Ericksonian Psychotherapy approach.The most important is the Garden of Revival which symbolizes the patient's health. It used to be full of life and energy, now it is neglected, requires work to be revived. In the therapeutic process day by day, the therapist tells the patient a symbolic story about his/her situation.
  Arms: VR Group
Behavioral: Cardiac rehabilitation — A three-week, hospital-based cardiac rehabilitation program for all participants, incorporating structured group exercises and activities. The conventional cardiac rehabilitation program includes morning warm-up exercises, afternoon group sessions, interval training on stationary bikes, and relaxation activities. Morning sessions consist of 20 minutes of standing cardiovascular exercises accompanied by music, while afternoon sessions include 45 minutes of seated activities, divided into cardiovascular, equipment-based, and breathing exercises.

SUMMARY:
The study aims to evaluate the effectiveness of virtual reality-assisted cardiac rehabilitation compared to conventional cardiac rehabilitation in improving psychological outcomes-depression, stress, anxiety, and kinesiophobia-along with physiological parameters, functional status, physical activity levels, and quality of life in cardiac patients.

DETAILED DESCRIPTION:
This single-blind randomized controlled trial will include 60 participants aged 60 years and older undergoing Phase II CR at the Provincial Specialist Hospital of the Blessed Virgin Mary in Częstochowa, Poland. Participants will be randomly assigned to one of two groups: a conventional CR program or a VR-CR group. Both groups will complete a three-week hospital-based CR program involving structured group exercises, interval cycling, and relaxation sessions. The experimental group will additionally receive eight sessions of immersive VR therapy using the VRTierOne device, consisting of 20-minute sessions twice weekly. These sessions employ interactive and calming virtual environments to promote relaxation and psychological engagement. Outcome measures will be evaluated at baseline (week 0), post-intervention (week 3), and follow-up (week 7). Assessments will include Patient-Reported Outcome Measures for stress, depression, kinesiophobia, and quality of life, physiological metrics (heart rate, blood pressure, metabolic equivalents), HRV, functional capacity (6MWT), and physical activity levels measured using the pedometers.

ELIGIBILITY:
Inclusion Criteria:

* cardiovascular diseases (atherosclerosis, hypertension, coronary artery disease, ischemic heart disease, peripheral artery disease, rheumatic heart disease, deep vein thrombosis, pulmonary embolism, and post-myocardial infraction)
* the second stage of cardiac rehabilitation conducted in outpatient settings

Exclusion Criteria:

* Severe psychiatric disorders (e.g., psychotic symptoms, bipolar disorder)
* initiation of psychiatric treatment or individual psychological therapy during the study period
* current use of antidepressant medications
* cognitive impairments that hinder questionnaire completion, consciousness disorders
* sensory impairments (e.g., severe visual or auditory deficits) that limit interaction with virtual reality.

Ages: 60 Months to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Tampa Scale for Kinesiophobia (TSK) at 3 and 7 weeks | From enrollment to the end of treatment at 3 weeks and follow-up at 7 weeks.
  TSK consists of 17 items designed to assess fear of movement and re-injury (kinesiophobia) in individuals experiencing pain or undergoing rehabilitation. Each item presents a statement regarding beliefs about movement and pain, with respondents indicating their level of agreement on a scale from 1 ("strongly disagree") to 4 ("strongly agree"). Total scores range from 17 to 68, with higher scores indicating greater levels of kinesiophobia. A score above 37 typically suggests a high degree of fear related to movement. Although the TSK primarily measures fear of movement, it can also indirectly reflect barriers to engagement in physical therapy.
Change from Baseline in the Short Form Health Survey (SF-36) at 3 and 7 weeks | From enrollment to the end of treatment at 3 weeks and follow-up at 7 weeks.
  SF-36 is a widely used 36-item questionnaire designed to assess health-related quality of life across various populations, including patients with chronic conditions. It evaluates eight domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional health, and mental health. Each domain is scored on a scale from 0 to 100, with higher scores indicating better health status and quality of life.
Change from Baseline in the Patient Health Questionnaire (PHQ-9) at 3 and 7 weeks | From enrollment to the end of treatment at 3 weeks and follow-up at 7 weeks.
  A nine-item instrument specifically designed for screening and assessing the severity of depression in primary care settings. Each item corresponds to a diagnostic criterion for major depressive disorder and asks respondents to reflect on their experiences over the past two weeks. Responses are scored on a scale from 0 ("not at all") to 3 ("nearly every day"), with total scores ranging from 0 to 27. Higher scores indicate more severe depressive symptoms, with scores of 5 or higher typically suggesting mild depression, and scores above 15 indicating moderate to severe depression.
Change from Baseline in the Exercise Capacity and Endurance at 3 and 7 weeks | From enrollment to the end of treatment at 3 weeks and follow-up at 7 weeks.
  The exercise conditions will be induced through a RAMP exercise test conducted on a treadmill, starting at a speed of 2.0 km/h with a 0% grade. Every 10 seconds, the speed and grade will increase incrementally by 0.1 to 0.15 km/h and 0.1% to 0.2%, respectively. To assess exercise capacity and endurance, metabolic equivalents (METs) will be calculated by determining the ratio of the metabolic work rate during exercise to the resting metabolic rate.

SECONDARY OUTCOMES:
Change from baseline in the autonomic nervous system activity at 3 and 7 weeks | From enrollment to the end of treatment at 3 weeks and follow-up at 7 weeks
  Autonomic nervous system activity will be assessed using heart rate variability (HRV), a measure that can serve as an indicator of psychological responses to stress. HRV will be recorded using the Polar H10 chest strap during a 5-minute measurement in a seated position. This method provides a reliable assessment of autonomic regulation, reflecting the balance between sympathetic and parasympathetic nervous system activity.
Change from Baseline in the Perceived Stress Scale (PSS-10) at 3 and 7 weeks | From enrollment to the end of treatment at 3 weeks and follow-up at 7 weeks.
  A tool for evaluating the level of perceived stress experienced by patients. This questionnaire consists of 10 items assessing various subjective feelings related to personal issues, life events, behaviors, and coping strategies over the past month. Respondents rate how often they have felt stressed or overwhelmed on a 5-point Likert scale, ranging from 0 ("never") to 4 ("very often"). Higher scores indicate greater levels of perceived stress, making it a valuable measure for understanding the impact of stress on patients' overall well-being.
Change from Baseline in the functional capacity at 3 and 7 weeks | From enrollment to the end of treatment at 3 weeks and follow-up at 7 weeks.
  Functional capacity will be assessed using the 6-Minute Walk Test (6MWT), which measures the distance a patient can walk in six minutes. This test provides valuable insights into exercise tolerance and overall physical ability. It is particularly effective for monitoring treatment efficacy, as improvements in walking distance often correlate with symptom relief and enhanced quality of life. The 6MWT is a submaximal exercise test that reflects the patient's functional capacity during daily activities, making it a practical and reliable measure, especially for individuals with moderate to severe cardiac or pulmonary conditions.
Daily physical activity levels during the rehabilitation period | From enrollment to the end of treatment at 3 weeks
  Physical activity levels will be assessed using a pedometer by recording step count with Yamax SW800-SW801 Digi-Walker Pedometer. The pedometer will be assigned to patients upon their qualification for the study, with instructions to use it throughout their entire stay.

CONTACTS AND LOCATIONS:
Overall Officials: Błażej Cieślik, PhD., Principal Investigator — Jan Dlugosz University in Czestochowa; Karolina Kowalewska, MSc., Principal Investigator — Jan Dlugosz University in Czestochowa
Locations (2):
- Poland (2):
  - Cardiac Rehabilita6on Department of the Provincial Specialist Hospital of the Blessed Virgin Mary in Czestochowa, Poland, Częstochowa, Upper Silesia
  - Jan Dlugosz University in Czestochowa, Częstochowa, Upper Silesia

IPD SHARING:
Plan to Share IPD: No